CLINICAL TRIAL: NCT07072026
Title: Feasibility of Endovascular Recanalization for Symptomatic Chronic Intradural Large Vessel Occlusions - Re-CHILL Study
Brief Title: Endovascular Recanalization for Symptomatic Chronic Intradural Occlusions
Acronym: Re-CHILL
Status: Recruiting | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-00410
Record Dates: First submitted 2025-06-16; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-06

CONDITIONS: Intracranial Stenosis; Intracranial Atherosclerotic Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background: Chronic intracranial large vessel occlusion (LVO), resulting from progressive atherosclerosis or thrombosis, contributes significantly to ischemic strokes, 8-10% in North America and up to 50% in the Chinese population. This condition leads to cerebral hypoperfusion, brain ischemia, and potentially cognitive impairment. While extra-to-intracranial bypass surgery has shown limited benefit, recent advances in endovascular treatment (EVT) for acute ischemic stroke show promise. Preliminary reports suggest EVT may be feasible for chronic intracranial artery occlusions. Still, outcomes vary and perioperative risks remain high, particularly for intradural occlusions, which are technically more challenging and less studied.

Objectives: This study aims to evaluate the feasibility, safety, and clinical outcomes of EVT for symptomatic chronic intradural large vessel occlusions. Primary endpoints include technical success, complication rates, and functional outcomes, as measured by the modified Rankin Scale (mRS) at 3 months and the last follow-up. Safety endpoints include mortality, ischemic stroke, and periprocedural complications.

Design: A multicenter, retrospective and prospective observational study involving 10-20 experienced centers worldwide. Data from approximately 40-80 patients treated between January 2020 and December 2024 will be collected by local neuroradiologists, neurologists, or neurosurgeons. Clinical data (demographics, comorbidities, symptoms, outcomes), imaging data (pre-, post-, and follow-up), procedural details, and medication regimens will be collected. Inclusion criteria target adult patients with symptomatic chronic intradural occlusions of key intracranial arteries (ICA, MCA, VA, BA). Symptomatic occlusion is defined by neurological deficits or imaging evidence of ischemia. The data analysis will be performed by the local team at the Inselspital, Bern, Switzerland.

Aim: To descriptively analyze patient characteristics, treatment approaches, complications, and hemodynamic changes post-EVT to inform future therapeutic strategies for this challenging condition.

ELIGIBILITY:
Inclusion Criteria:

* all consecutive patients who undergone endovascular recanalization for chronic intradural large vessel occlusions between January 1st, 2020, and December 31st, 2024 involving the following locations: internal carotid artery (ICA), middle cerebral artery (MCA), vertebral artery (VA), and basilar artery (BA)

Exclusion Criteria:

* presence of documented written or verbal refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The intradural occlusion is defined as the occlusion entirely located or extended into an intradural vascular segment (e.g., ICA occlusion extending from the extradural ICA to the ophthalmic ICA segment).
  The ICA segments are defined as follows:
  * Extradural ICA segment - from the ICA origin until the distal dural ring
  * Ophthalmic ICA segment - from the distal dural ring right below the origin of the posterior communicating artery (PCOM)
  * Communicating ICA segment - right from the PCOM origin to the ICA termination (bifurcation)
  The symptomatic occlusion is defined as acute neurological impairment and/or acute ischemic stroke or hypoperfusion within the affected vascular territory detected on baseline imaging.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical outcome assesed by modified Rankin Scale | at 3 months after endovascular treatment
  The primary outcome is the degree of dependency and disability in everyday life measured with the modified Rankin Score (mRS) at 90 days. The mRS is the standard tool to assess neurological outcome in trials with acute severe brain disease. The scale runs from 0-6, running from perfect health without symptoms (= 0) to death (= 6).
Rate of technical success | on the day of procedure
  Succesful versus failed recanalization; presence or absence of the residual stenosis

SECONDARY OUTCOMES:
Clinical outcome at the last available follow-up assesssed by modified Rankin Score | through study completion, an average of 1 year
  Degree of dependency and disability in everyday life measured with the modified Rankin Score (mRS) . The mRS is the standard tool to assess neurological outcome in trials with acute severe brain disease. The scale runs from 0-6, running from perfect health without symptoms (= 0) to death (= 6).
Death during the initial hospital stay | from day 1 until discharge from hospital, on average of 7 days
Death at 3 months | from day 1 up to 3 months
  occurence of death from day 1 up to 3 months

OTHER OUTCOMES:
New Ischemic stroke on the follow-up imaging | from the day of treatment through study completion, an average of 6 months
  Radiologic occurrence of newly evolved ischemic stroke (hypodenisty or parenchymal defect on computer tomographie scan, or hyperintense lesion on T2 weighted/fluid-attenuated inversion recovery scan with or without corresponding restricted diffusion)
Rate of periprocedural and postprocedutral complications | from the endovascular treatment through study completion, an average of 6 months
  Any periprocedura complications including vessel perforation, acute in-stent thrombosis, distal thromboembolisation, complication in the access site (hematoma in situ, retroperitoneal hematoma, pseudoaneurysma, etc.). Detection of asymptomatic or symptomatic in-stent thrombosis or in-stent stenosis on follow-up angiography scan (computer tomographie angiography, magnetic resonance angiography, or digital subtraction angiography).

CONTACTS AND LOCATIONS:
Locations (2):
- Alfried Krupp Krankenhaus, Essen, Germany
- Inselspital Bern, University Hospital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No